CLINICAL TRIAL: NCT01822964
Title: Oxygenation of the Cerebrum and Cooling During Transcatheter Aortic Valve Implantation (TAVI) Procedures - Part II
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Prof Dr Cathy De Deyne, Prof Dr, dept of physiology, Hasselt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OCCTAVI-II; TAVI research funding (Other: Hasselt University)
Record Dates: First submitted 2013-03-24; First posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-03

CONDITIONS: Aortic Valve Stenosis; Stroke
MeSH Terms: conditions — Aortic Valve Stenosis; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- targeted brain cooling (Active Comparator): In these 15 pts, targeted brain cooling (tympanic temperature of 33°C) will be applied during the TAVI intervention by the use of the RhinoChill device (Benechill Inc, San Diego cA)
  Interventions: Device: targeted brain cooling (33°C) by RhinoChill device
- no use of targeted brain cooling (Placebo Comparator): In these 15 pts, no cooling techniques will be applied and current clinical practice as to maintenance of normothermia will be followed during these TAVI interventions
  Interventions: Device: Placebo - current clinical practice, no cooling

INTERVENTIONS:
Device: targeted brain cooling (33°C) by RhinoChill device — targeted brain cooling by Rhinochill device to 33°C tympanic temperature during TAVI procedure. After valve implantation, slow rewarming until 35.5°C
  Arms: targeted brain cooling
Device: Placebo - current clinical practice, no cooling
  Arms: no use of targeted brain cooling

SUMMARY:
The aim of this study is to assess the possible neuroprotective effects of cooling (targeted cooling of the brain to 33°C) during Transcatheter Aortic Valve Implantation (TAVI) procedures. From start of anesthesia, until final valve implantation, local cooling (by the RhinoChill device) will be applied to the brain. Effect of cooling on cerebral oxygenation, by cerebral oxygen saturation monitoring (NIRS ForeSight technology) during the TAVI procedure will be continuously assessed during native valve manipulation and during final valve deployment (=primary endpoint of he study). As secondary endpoints, neuropsychological testing performed before and after TAVI procedure will assess the effects of the use of cooling during the TAVI procedure. Neuron-specific enolase (NSE) and S100-beta will be analyzed during and up to 72hrs after TAVI to compare the cerebral ischemic damage between cooled and non-cooled patients. And finally, diffusion-weighted MRI of the brain will be performed 5 days before and 5-7 days after TAVI to compare the number and total amount of cerebral ischemic insults between cooled and non-cooled patients. The hypothesis behind this study is that by local cooling of the brain during manipulation of the calcified aorta and aortic valve, the brain might be protected from cerebral ischemic insults.

ELIGIBILITY:
Inclusion Criteria:

* pts scheduled for transcatheter aortic valve implantation

Exclusion Criteria:

* pts with pacemaker already implanted
* pts with recent stroke or Transient Ischemic Attacks (TIA) (6months)
* pts with extreme claustrophobia for MRI brain examination

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
changes in cerebral oxygen saturation during periods of rapid ventricular pacing and valve implantation | during TAVI procedure
  changes in cerebral oxygen saturation during periods of rapid ventricular pacing (RVP) and valve implantation; changes in cerebral oxygen saturation compared to baseline values (of 10min) before periods of RVP (Area Under the Curve will be analysed and compared between cooled end non-cooled patients

SECONDARY OUTCOMES:
composite outcome measure : MRI of the brain before and after TAVI; NSE before and after TAVI; S100-B before and after TAVI; neuropsychological testing before and after TAVI | one year

OTHER OUTCOMES:
composite outcome measure : General Clinical Endpoints (as referring to the Valval Academic Research Consortium (VARC) - 2 recommendations) | one year
  These clinical endpoints include : all-cause mortality; myocardial infarction; stroke & TIA; bleeding complication; acute kidney injury; vascular complications; conductance disturbances and arrhythmias; other TAVI-related complications; valvular function and quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Cathy S De Deyne, Md, PhD, Principal Investigator — University Hasselt / Ziekenhuis Oost-Limburg Genk (Belgium)
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - Universitair Ziekenhuis, Leuven

REFERENCES:
- [Background] 1. Vahanian A, Alfieri O, Al-Attar N, Antunes M, Bax J, Cornier B, Cribier A, De Jaegere P, Fournial G, Kappetein AP et al. Transcatheter valve implantation for patients with aortic stenosis: a position statement from the European association of cardio-thoracic surgery (EACTS- and the European Society of Cardiology (ESC), in collaboration with the European Association of Percutaneous Cardiovascular Interventions (EAPCI). Eurointervention 2008;4:193-199 2. Leon MB, Smith CR, Mack M, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR et al. Transcatheter aortic-valve implantation for aortic stenosis in patients who cannot undergo surgery. N Eng J Med 2010;363:1597-1607 3. Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tizcu EM, Webb JG, Fontana GP, Makkar RR et al. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Eng J Med 2011;364:2187-2198 4. Grube E, Naber C, Abizaid A, Sousa E, Mendiz O, Lemos P et al. Feasibility of transcatheter aortic valve implantation withoutn balloon pre-dilatation. JACC Cardiovasc Interv 2011;4:751-757 5. Bagur R, Rodes-Cabau J, Doyle D, De Larochelière R, Villeneuve J, Bertrand OF et al. Transcatheter aortic valve implantation with